CLINICAL TRIAL: NCT03021512
Title: Retrospective Functional Assessment of Activities of Daily Living (ADL) in Patients Who Underwent Bilateral Implantation of Aspheric Bifocal Intraocular Lenses or Aspheric Trifocal Intraocular Lenses
Brief Title: Functional Assessment of ADL in Patients Who Underwent Bifocal and Trifocal Presbyopic Correction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Assistant Professor, Democritus University of Thrace
Other Study IDs: 299/13-1-2017
Record Dates: First submitted 2017-01-13; First posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1 (BFG): (Bifocal group). Subjects that underwent bifocal intraocular lenses implantation. (ie. Phaco with Restor intervention).
  Interventions: Procedure: Phaco with Restor
- Group 2 (TFG): (Trifocal group). Subjects that underwent trifocal intraocular lenses implantation. (ie. Phaco with Panoptix intervention).
  Interventions: Procedure: Phaco with Panoptix

INTERVENTIONS:
Procedure: Phaco with Restor — Phacoemulsification with bilateral bifocal intraocular lenses implantation
  Groups: Group 1 (BFG)
Procedure: Phaco with Panoptix — Phacoemulsification with bilateral trifocal intraocular lenses implantation
  Groups: Group 2 (TFG)

SUMMARY:
Patients who underwent bilateral bifocal or trifocal lenses implantation for presbyopia correction with monofocal intraocular lenses implantation are supposed to have sufficient uncorrected vision capacity for activities of daily living (ADLs) that require: a) distant vision (DV), (ie. driving), b) intermediate vision (IV), (ie. computer word processing), c) near vision (NV), (ie. book reading). Primary objective of the study is the comparison in a series of ADLs of two cohorts of patients (group 1: subjects with bilateral bifocal lenses implantation, group 2: subjects with bilateral trifocal lenses implantation)

ELIGIBILITY:
Inclusion Criteria:

* Presbyopic patients that underwent either bilateral bifocal or trifocal intraocular lenses implantation

Exclusion Criteria:

* Glaucoma, Corneal pathology, Fundus pathology, Mental or Neurological disorder

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Grade 1 Cataract Patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Visual Capacity (VC) | 1 year following surgery
  Assessment of Visual capacity (VC)

SECONDARY OUTCOMES:
Distant Visual Capacity (DVC) | 1 year following surgery
  Visual capacity for activities that require distant vision (DVC). DVC score will be measured by the performance score in the following ADLs: a) walking specific pathway, 2) walking up stairs, 3) walking down stairs, 4) day-time driving simulation, 5) night-time driving simulation
Intermediate Visual Capacity (IVC) | 1 year following surgery
  Visual Capacity for activities that require intermediate vision (IVC). VC score will be measured by the performance score in the following ADLs: a) reading ability of movie subtitles, b) reading ability of a predefined computer screen text, c) reading a supermarket badge
Near Visual Capacity (NVC) | 1 year follwoing surgery
  Visual Capacity for activities that require near vision (NVC). NVC score will be measured by the performance score in the following ADLs: a) cellular phone directory entry search, b) reading of message in a cellular phone, c) reading a medical prescription, d) reading a public phonebook

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Democritus University of Thrace, Alexandroupoli, Evros, Greece

IPD SHARING:
Plan to Share IPD: No